CLINICAL TRIAL: NCT05672069
Title: Ambispective, Multicentre, Open-label Study Evaluating the Clinical Outcomes of Foot Surgery Using SERF Medical Devices
Status: Completed | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-08
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-04

CONDITIONS: Foot Diseases
MeSH Terms: conditions — Foot Diseases | interventions — Fracture Fixation, Internal; Arthrodesis; Osteotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Osteosynthesis — Foot pathologies
  Other Names: Arthrodesis; Osteotomy

SUMMARY:
This clinical investigation was led as a post-marketing clinical follow-up study conducted as part of standard care with an additional, non-invasive, non-invasive procedure (Case 4.1) ambispective, multicentre, open-label, non-comparative.

The primary objective of this study is to evaluate the reduction in patient pain and the restoration of walking. The study will also collect performance and safety data to assess the subject's outcomes and functional status.

The target population for this study was any adult patient implanted with FAST screws, FAST plates, Toe FAST and VEOFIX screws between november 2021 and october 2022.

The investigation will be conducted in accordance with the investigation protocol, the laws and regulations (including the Medical regulations (including the Medical Devices Regulation 2017/745) and the ISO 14155:2020, as well as in accordance with the ethical principles described in the Declaration of Helsinki. The collection of personal data will also be compliant with RGPD 2016/679.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of legal age at the date of implantation;
* Subject implanted with one or more implants: FAST Screw, FAST Plate, Toe FAST and VEOFIX Screw between November 2021 and October 2022;
* Subject able to understand the information and instructions given by the investigator;
* Subject with a social security affiliation.

Exclusion Criteria:

* Vulnerable persons
* People with contraindications (including pregnant women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women of legal age, for whom one of the devices is implanted according to the instructions for use. These patients will be monitored according to standard care. As the series is observational and has an additional procedure that is neither burdensome nor invasive, all implanted patients will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Saint-Martin, Pessac, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Cohort: The description will be carried out on the whole population really included
Period: Overall Study
Arm/Group | Total Cohort
Started | 124
Completed | 121
Not Completed | 3
Not completed — Implant removal | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Total Cohort
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.20 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  French nationality | 124
Operated foot side [Number; unit: Number of foot]
  Right | 65
  Left | 72
Foot position [Number; unit: Number of foot]
  Front of foot | 123
  Middle of foot | 6
  Front + Middle of foot | 3
  Back of foot | 5
Weight (kg) [Mean (Standard Deviation); unit: Kg] | 66.72 (14.12)
Height of participant (cm) [Mean (Standard Deviation); unit: cm] | 165.85 (7.23)

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Patient's Pain and Restoration of Walking
Description: The information will be collected through AOFAS (American Orthopaedic Foot and Ankle Society) score (>80 points) at 12 months. This score is assessed using a questionnaire measuring the patient's pain, function and alignment of the foot. This score range from 0 (worst score) to 100 (best score). The score is interpreted as follows :
  Between 90-100 points : excellent results Between 80-89 points : good results Between 60-79 points : fair results Less than 60 points : poor results This score is composed of 3 sub-scores : (i) Pain score is ranging from 0 to 40 points ; Function score is ranging from 0 to 45 points ; Alignment is ranging from 0 to 15 points.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Total Cohort
Number analyzed (Participants) | 121
points
  Preoperatively | 42.46 (15.25)
  12 months | 88.44 (13.50)

2. Secondary Outcome: Survival Rate
Description: Determination of the Kaplan-Meier type survival curve, with any revision as the endpoint whatever the cause. At each inflection point, a revision surgery with removal or revision surgery with removal or change of a component of the implant under consideration All causes of revision are considered. Patients who have died or been lost to follow-up will be included in the analysis.
Time Frame: 12 months
Measure: Number; unit: percentage of implant survivorship
Arm/Group | Total Cohort
Number analyzed (Participants) | 121
percentage of implant survivorship | 89.3

3. Secondary Outcome: Foot Bone Consolidation
Description: The information will be collected through investigator's question : "on radiographic reading, is the foot bone consolidation satisfactory? : 4 answers are proposed: "total / partial / null / no information".
Time Frame: 12 months
Measure: Number; unit: Number of foot
Arm/Group | Total Cohort
Number analyzed (Participants) | 121
Number of foot
  Total | 124
  Partial | 2
  No consolidation | 1
  Not determined | 7

4. Secondary Outcome: Patient Satisfaction
Description: The information will be collected through patient's question : "Considering your expectations, are you satisfied with your operation?" 4 answers are proposed: "I am completely satisfied with the results of my operation results of my operation / My condition has not improved as much as I had hoped, but I but I would be willing to have the same operation for the same result / The operation improved my condition, but I would not be prepared to have the same operation for the same result / My condition is the same or worse than before my operation than before my operation".
Time Frame: 12 months
Measure: Number; unit: Number of foot
Arm/Group | Total Cohort
Number analyzed (Participants) | 121
Number of foot
  Very satisfied | 103
  Satisfied | 20
  Neither satisfied nor unsatisfied | 6
  Unsatisfied | 5

5. Secondary Outcome: Adverse Event
Description: Type and occurrence of adverse events
Time Frame: Peroperative to 12 months
Measure: Number; unit: Number of foot
Arm/Group | Total Cohort
Number analyzed (Participants) | 121
Number of foot
  Discomfort | 8
  Pain | 3
  Pseudoarthrosis | 2
  Screw protrusion | 2
  Persistent pain (consolidation with screw protrusion) | 1
  Post-operative neurological disorders | 1
  Stiff joint (hallux positioning problem) | 1
  Loss of correction | 1
  Scar disunion (poor effectiveness of meching) | 1
  Locking default between locking screws/plate | 1

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Total Cohort: The adverse event occurred in an implanted foot.
Arm/Group | Total Cohort
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 5/121
Other Adverse Events (participants affected / at risk) | 16/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Cohort (N=121)
Persistent pain (consolidation with screw protrusion) (Surgical and medical procedures) | 1
Arthrodesis pseudarthrosis (Surgical and medical procedures) | 1
Post-operative neurological disorders (Nervous system disorders) | 1
Screw protrusion (Surgical and medical procedures) | 1
Pseudarthrosis (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Cohort (N=121)
Persistent / residual pain (Injury, poisoning and procedural complications) | 3
Screws protrusion (Surgical and medical procedures) | 1
Discomfort (Injury, poisoning and procedural complications) | 8
Loss of correction (Surgical and medical procedures) | 1
Scar disunion (poor effectiveness of meching) (Surgical and medical procedures) | 1
Locking default between locking screws /plate (Surgical and medical procedures) | 1
Stiff joint (hallux positioning problem) (Surgical and medical procedures) | 1

LIMITATIONS AND CAVEATS:
This investigation had planned to collect 320 patients (40 per surgeon). However, the amount of data collected for FAST plates (and associated screws), VEOFIX screws and Toe FAST is limited due to a lack of inclusion or an overestimation of the capacity of the investigation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT05672069/Prot_000.pdf